CLINICAL TRIAL: NCT03193931
Title: A Randomized Phase II Study Comparing Pembrolizumab With Methotrexate in Elderly, Frail or Cisplatin-ineligible Patients With Head and Neck Cancers
Brief Title: Study Comparing Pembrolizumab With Methotrexate in Elderly, Frail or Cisplatin-ineligible Patients With Head and Neck Cancers
Acronym: ELDORANDO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: A very low recruitment rate made it impossible to reach the recruitment goal wthin an acceptable timeframe.
Sponsor: AIO-Studien-gGmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO-KHT-0115
Record Dates: First submitted 2017-05-31; First posted 2017-06-21 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Cancer of Head and Neck
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Patients recieve pembrolizumab or methotrexate
Masking Description: opern label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Pembrolizumab 200 mg q3w i.v. until disease progression or non-tolerable toxicity (maximum 2 years)
  Interventions: Drug: Pembrolizumab Injection
- Arm B (Active Comparator): Arm B: Methotrexate (MTX) 40 mg/m2 weekly i.v. until disease progression or non-tolerable toxicity (maximum 2 years)
  Interventions: Drug: Methotrexate Injectable Solution

INTERVENTIONS:
Drug: Pembrolizumab Injection — Pembrolizumab 200 mg q3w i.v. until disease progression or non-tolerable toxicity (maximum 2 years)
  Arms: Arm A
Drug: Methotrexate Injectable Solution — Methotrexate 40 mg/m2 weekly i.v. until disease progression or non-tolerable toxicity (maximum 2 years)
  Arms: Arm B

SUMMARY:
The study is designed as an open-label, randomized, prospective, multicenter, phase II study comparing pembrolizumab with methotrexate in elderly, frail or cisplatin-ineligible patients with squamous carcinoma of the head and neck (HNSCC)

ELIGIBILITY:
Inclusion Criteria:

1. Cooperation and willingness to complete all aspects of the study
2. Signed written informed consent must be given prior to study inclusion
3. Histological or cytological confirmed recurrent or metastatic squamous cell carcinoma of the head and neck (HNSCC) not amenable to local therapies
4. Progressive disease at study entry
5. At least 1 measurable lesion according to RECIST 1.1
6. No previous systemic treatment for metastatic disease
7. Not eligible for cisplatin-based chemotherapy, defined as:

   * ECOG 2 [Eastern Cooperative Oncology Group] and/or
   * Calculated CrCl [Creatinine Clearance] <60 mL/min (measured by MDRD)
8. Age ≥ 18 years
9. ECOG performance status 0 - 2
10. Brain metastases require completion of local therapy with discontinuation of steroids prior to start of treatment
11. If of childbearing potential, willingness to use highly effective contraceptive method for the duration of the study and 120 days after last dose, such as combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), vasectomized partner, bilateral tubal occlusion, sexual abstinence. If an oral contraception is used, a barrier method of contraception (e.g. male condom, female condom, cervical cap, diaphragm, contraceptive sponge) has to be applied additionally.
12. Adequate bone marrow function, liver and renal function:

    1. Absolute neutrophil count ≥ 1.5 x 109/L
    2. Thrombocytes ≥ 100 x 109/L
    3. Hemoglobin ≥ 9 g/dL
    4. INR [international normalized ratio] ≤ 1.5 and PPT [partial prothrombin time] ≤ 1.5 x lower limit during the last 7 days before therapy
    5. Bilirubin < 1.5 x lower limit and
    6. AST (GOT) [aspartate aminotransferase] and ALT (GPT) [alanine transaminase] < 3 x lower limit (5 x lower limit in case of liver metastases)
13. Tumor block or 20 slides must be available at study inclusion for central pathology testing

Exclusion Criteria:

1. Live expectancy less than 3 months
2. Nasopharynx carcinoma
3. Anticancer treatment during the last 30 days prior to start of treatment, including systemic therapy, radiotherapy or major surgery
4. Participation in a clinical trial within the last 30 days prior to study treatment
5. History of allogeneic tissue/solid organ transplant
6. History of pneumonitis that has required oral or i.v. steroids
7. Evidence of interstitial lung disease
8. Minor surgery ≤ 24 hours prior first dose of study treatment
9. Symptomatic acute cardiovascular or cerebrovascular disease
10. Known active HBV [hepatitis B virus], HCV [hepatitis C virus] or HIV infection
11. Has any other active infection requiring systemic therapy.
12. Patients with active tuberculosis
13. Prior therapy with an anti-Programmed cell death protein 1 (anti-PD-1), anti-PD-L1, anti-Programmed cell death-ligand 2 (anti-PD-L2), anti-CD137 (4-1BB ligand, a member of the Tumor Necrosis Factor Receptor (TNFR) family), or anti-Cytotoxic T-lymphocyte-associated antigen-4 (anti-CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
14. A diagnosis of immunodeficiency or patient is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
15. Patient has had a prior monoclonal antibody, which does significantly interfere with the immune system or which does have a systemic therapeutic effect on the tumor within 4 weeks prior to randomization.
16. Patient has not recovered (i.e., ≤ Grade 1 or at baseline) from any toxicity due to agents administered more than 4 weeks earlier. [Subjects with ≤ Grade 2 neuropathy or alopecia are an exception to this criterion and may qualify for the study.]
17. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
18. Has received a live vaccine within 30 days prior to the first dose of trial treatment.
19. Has known hypersensitivity to methotrexate or pembrolizumab or any constituent of the products..
20. Other active malignancy requiring treatment
21. Lactating or pregnant women, women of child-bearing potential who do not agree to the usage of highly effective contraception methods (allowed methods of contraception, meaning methods with a rate of failure of less than 1% per year are combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), vasectomized partner, bilateral tubal occlusion, sexual abstinence. If an oral contraception is used, a barrier method of contraception (e.g. male condom, female condom, cervical cap, diaphragm, contraceptive sponge) has to be applied additionally). Women of childbearing potential must have a negative pregnancy test (serum β-hCG) at Screening.
22. Any psychiatric illness that would affect the patient's ability to understand the demands of the clinical trial
23. Patient has already been recruited in this trial (does not include screening failures)
24. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities § 40 Abs. 1 S. 3 Nr. 4 AMG.
25. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
Antitumor activity of pembrolizumab in SCCHN | 1 year
  Overall survival (OS) rate

SECONDARY OUTCOMES:
Quality of life QLQC30 [EORTC QLQ-C30] | through study completion, an average of 6 years
  QLQC30
Quality of life HN35 [EORTCQLQ-H&N35] | through study completion, an average of 6 years
  HN35
Predictive biomarkers | through study completion, an average of 6 years
  molecular-genetic pro-inflammatory markers
Predictive biomarkers | through study completion, an average of 6 years
  PD-L1 expression
Time to failure of strategy (TTFS) | 1 year
  defined as death, progressive disease (PD), treatment discontinuation ( or deterioration of Instrumental Activities of Daily Living (IADL score) by 2 points.
Efficacy of pembrolizumab in SCCHN | through study completion, an average of 6 years
  Objective response rate (ORR) according to RECIST 1.1
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | through study completion, an average of 6 years
  Adverse event rates due to treatment with MTX and pembrolizumab in SCCHN measured according to CTCAE 4.03

OTHER OUTCOMES:
QoL response QLQC30 | through study completion, an average of 6 years
  improvement in QLQC30
QoL response HN35 | through study completion, an average of 6 years
  improvement in HN35
prognostic value of tumor shrinkage | through study completion, an average of 6 years
  objective response rate (ORR) according to RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Medizinsche Hochschule Hannover, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No